CLINICAL TRIAL: NCT03401346
Title: A Phase I, Three-Period, Three-Way, Randomized, Open-Label, Single-Dose, Cross-Over, Comparative Bioavailability Study of Dihydroergotamine Mesylate (DHE) Administered by I123 Precision Olfactory Delivery (POD) Device Nasal Spray, DHE for Injection (Intravenous), and Migranal® Nasal Spray in Healthy Adult Subjects
Brief Title: Bioavailability of DHE Administered by I123 POD Device, IV Injection, and Migranal Nasal Spray in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INP104-101; ACTRN12617001381370p (Registry Identifier: ANZCTR)
Record Dates: First submitted 2017-12-17; First posted 2018-01-17 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-01

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- INP104 (Experimental): Single dose 1.45 mg Dihydroergotamine Mesylate (DHE), administered by I123 Precision Olfactory Delivery (POD) device nasal spray (INP104)
  Interventions: Combination Product: INP104
- D.H.E. 45 Injection (IV) (Active Comparator): Single dose 1 mg Dihydroergotamine Mesylate (DHE) for intravenous injection
  Interventions: Drug: Dihydroergotamine Mesylate (DHE)
- Migranal Nasal Spray (Active Comparator): Single dose 2 mg Migranal Nasal Spray Dihydroergotamine Mesylate (DHE)
  Interventions: Combination Product: Migranal Nasal Spray

INTERVENTIONS:
Combination Product: INP104 — Dihydroergotamine Mesylate (DHE) administered via I123 Precision Olfactory Delivery (POD) Device
  Arms: INP104
Drug: Dihydroergotamine Mesylate (DHE) — Dihydroergotamine Mesylate (DHE) injection (intravenous)
  Arms: D.H.E. 45 Injection (IV)
Combination Product: Migranal Nasal Spray — Dihydroergotamine Mesylate (DHE) delivered via Migranal Nasal Spray pump
  Arms: Migranal Nasal Spray

SUMMARY:
A Phase I clinical trial to compare the bioavailability of dihydroergotamine mesylate (DHE) following a single dose administration of INP104 (DHE administered by I123 Precision Olfactory Delivery (POD) Device Nasal Spray) to that of D.H.E. 45 for Injection (Intravenous) and Migranal Nasal Spray in healthy adult subjects.

It is hypothesized that INP104 will address the current variability in nasal administration and give more reproducible dose delivery compared to Migranal nasal spray.

Blood concentrations of all three investigational products will be compared for 48 hours following dosing. The safety and tolerability of INP104 will be monitored throughout the study.

INP104 has been developed for the treatment of acute migraine headache. The device in which the drug will be delivered has been designed to deliver the medication to the upper nasal cavity with minimal variation in dose absorption, eg loss via dripping out of the nose or the dose being swallowed.

Approximately 36 participants in general good health (equal ratio of males and females desired) will be enrolled and will be allocated to receive 3 treatments in a randomized sequence. They will receive a single dose of INP104, a single dose of DHE via intravenous injection, and a single dose of Migranal Nasal Spray. There will be a wash out period where no treatment will be administered for 7 days in between each treatment. Participants are required to attend 3 inpatient periods and 1 final outpatient visit. Each participant will be in the study for up to 43 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females, 18 to 55 years of age (inclusive) at the time of screening.
* Subjects must be in good general health, with no significant medical history (including migraine), have no clinically significant abnormalities on physical examination at screening, and/or before administration of the initial dose of investigational product.
* Subjects must have a Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive.
* Subjects must have clinical laboratory values within normal range as specified by the testing laboratory, or assessed as not clinically significant by the Principal Investigator.
* Negative urine drug screen/alcohol breath test at screening.
* Subjects who are willing to refrain from smoking for the duration of the study.

Exclusion Criteria:

* Subjects with a recent history of migraine and its variants including hemiplegic migraine and basilar migraine. A recent history of migraine is defined as (a) current or past history of migraine with at least 1 attack in last 6 months or (b) those receiving antimigraine prophylaxis.
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
* Subjects who have ingested caffeine within 48 hours before admission on Day -1. Subjects must also agree to refrain from consumption of caffeinated drinks for 48 hours before admission of Days 7 and 14 (i.e. prior to each subsequent dosing), and throughout confinement.
* Subjects with ischemic heart disease or subjects who have clinical symptoms or findings consistent with coronary artery vasospasm including Prinzmetal's variant angina.
* Subjects with hypertension, known peripheral arterial disease, Raynaud's phenomenon, sepsis, history of vascular surgery or severely impaired hepatic or renal function
* Subjects who have previously shown hypersensitivity to ergot alkaloids or metoclopramide.
* Use of any relevant prescription, over-the-counter medication (with the exception of oral contraceptives), foods (e.g. grapefruit juice) or supplements (including herbal) within 14 days of randomization [especially those affecting the Cytochrome P450 3A4 (CYP3A4) metabolic pathway].
* History or presence of alcoholism or drug abuse within the 2 years prior to the first investigational product administration.
* Surgery within the past three months prior to the first investigational product administration as determined by the PI to be clinically relevant.
* Active infection and/or use of macrolide antibiotics within 14 days prior to enrollment.
* History of recurrent infections.
* Any nasal congestion or physical blockage in either nostril, or deviated nasal septum as determined by nasal examination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
DHE pharmacokinetics | 48 hours
  Cmax
DHE pharmacokinetics | 48 hours
  Tmax
DHE pharmacokinetics | 48 hours
  AUC(0-t)
DHE pharmacokinetics | 48 hours
  kel
DHE pharmacokinetics | 48 hours
  T(1/2)
DHE pharmacokinetics | 48 hours
  AUC(0-inf)
DHE pharmacokinetics | 48 hours
  CL/F (CL for IV administration)

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 1 to day 22 post first dosing
  Incidence of treatment-emergent adverse events after one dose of INP-104, Migranal Nasal Spray or DHE45 by IV injection
8'-OH-DHE pharmacokinetics | 48 hours
  Cmax
8'-OH-DHE pharmacokinetics | 48 hours
  Tmax
8'-OH-DHE pharmacokinetics | 48 hours
  AUC(0-t)
8'-OH-DHE pharmacokinetics | 48 hours
  kel
8'-OH-DHE pharmacokinetics | 48 hours
  T(1/2)
8'-OH-DHE pharmacokinetics | 48 hours
  AUC(0-inf)
8'-OH-DHE pharmacokinetics | 48 hours
  CL/F (CL for IV administration)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Centre for Clinical Studies/Nucleus Network
Locations (1):
- Centre for Clinical Studies/Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shrewsbury SB, Jeleva M, Satterly KH, Lickliter J, Hoekman J. STOP 101: A Phase 1, Randomized, Open-Label, Comparative Bioavailability Study of INP104, Dihydroergotamine Mesylate (DHE) Administered Intranasally by a I123 Precision Olfactory Delivery (POD(R) ) Device, in Healthy Adult Subjects. Headache. 2019 Mar;59(3):394-409. doi: 10.1111/head.13476. Epub 2019 Jan 19. PMID 30659611